CLINICAL TRIAL: NCT02157766
Title: Wisconsin Center for the Neuroscience and Psychophysiology of Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-0116; P01AT004952 (NIH)
Record Dates: First submitted 2014-05-27; First posted 2014-06-06 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2019-05

CONDITIONS: Mindfulness; Compassion; Meditation; Mental Health; Asthma
Keywords: Mental Health; Asthma; Mindfulness; Compassion; Meditation
MeSH Terms: conditions — Psychological Well-Being; Asthma | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MNP with Asthma: Mindfulness Based Stress Reduction (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- MNP w/ Asthma: Wait List Control (No Intervention)
- MNP, no asthma - Mindfulness Based Stress Reduction (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- MNP, no asthma: Health Enhancement Program (Active Comparator)
  Interventions: Behavioral: Health Enhancement Program
- MNP, no asthma - Wait List Control (No Intervention)
- Long Term Meditator (Active Comparator)
  Interventions: Behavioral: Intensive Meditation Practice

INTERVENTIONS:
Behavioral: Intensive Meditation Practice — Long term meditators complete three days of of mindfulness or compassion/loving kindness meditation at T2 and T3 (one meditation type per visit).
  Arms: Long Term Meditator
Behavioral: Mindfulness Based Stress Reduction — 8 week class designed to enhance well-being through training in mindfulness.
  Other Names: MBSR
  Arms: MNP with Asthma: Mindfulness Based Stress Reduction; MNP, no asthma - Mindfulness Based Stress Reduction
Behavioral: Health Enhancement Program — 8 week class designed to enhance well-being through training in physical activity, functional movement, music therapy and nutrition.
  Other Names: HEP
  Arms: MNP, no asthma: Health Enhancement Program

SUMMARY:
The Wisconsin Center for the Neuroscience and Psychophysiology of Meditation will be a highly focused center dedicated to novel and cutting edge research on the mechanisms by which meditation works. The core set of hypotheses for this Center focus on the mechanisms of two common meditation practices: Mindfulness Meditation (MM) and Loving-Kindness/Compassion Meditation (LKM-CO), both taught in Mindfulness-Based Stress Reduction (MBSR). The investigators will study both Long-Term Meditators (LTMs) as well as meditation-naïve participants (MNPs). The latter group will be randomly assigned to MBSR, a rigorously matched comparison intervention called the Health Enhancement Program (HEP; MacCoon et al., 2012), or to a Wait List (WL) control group. This will give us a comprehensive view of changes that are produced by meditation practices per se, changes generically associated with interventions designed to promote well-being, and changes that might be effects of repeating testing protocols across multiple occasions. In addition, the inclusion of both novice and experienced meditators provides a wide range of practice experience that will provide critical information on dose-related effects, information that is lacking in the research literature today.

Each of the projects is focused on examining the brain mechanisms and peripheral biological correlates of meditation. Project 1 (Davidson) will examine the impact of the explicit use of mindfulness and loving-kindness/compassion strategies on emotion regulation, specifically neural, biobehavioral and hormonal indices of reactivity to and recovery from pictures of human suffering and flourishing. Project 2 (Rosenkranz) will investigate the brain to periphery pathways through which psychological factors contribute to the expression of asthma symptoms. In addition, it will examine the efficacy of meditation training in reducing the inflammatory response to an allergen in asthmatic individuals by reducing the reactivity of emotion-related neural circuitry. Project 3 (Tononi) will examine whether the previously reported increase in gamma oscillations during Non-REM (NREM) sleep in meditators is associated with changes in sleep mentation (Ferrarelli et al. 2013). In addition, project 3 will examine relations between meditation-induced changes in brain activity during sleep and brain activity and cognitive function during wakefulness.

ELIGIBILITY:
Inclusion Criteria - MNP-A:

* Able to provide valid informed consent to participate by signing/dating a consent form.
* Fluent English speaker
* MRI safe - Not excluded based on magnetic resonance Screening Form
* 18-65 years old
* Pre-albuterol FEV1 ≥ 60% while holding meds
* Physician's diagnosis of asthma - via clinical assessment, reversibility or airway hyperresponsivity;
* Ability to provide blood samples with relatively easy vascular access
* Uses acceptable contraception
* Evidence of persistent, residual inflammation (≥2% sputum eosinophils OR peripheral blood eosinophils ≥ 150 OR eNO of 30+
* Must be US citizen, green card holder or have an F-1 or J-1 visa. This is required in order to be able to pay participants.

Exclusion Criteria - MNP-A:

* Pregnant, wanting to become pregnant, breast feeding or less than 6 months post-partum.
* Taking prescribed psychotropic or central nervous system altering medications (may be included with the PIs discretion).
* History of a diagnosed Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder. Diagnosed episode of Major Depression unless it was more than 1 year ago. Diagnosed eating disorder or anxiety disorder unless it was more than 1 year ago. (May be included with the PIs discretion).
* Excluded based upon the screening visit
* Some ongoing medical problems will be excluded based on team judgments about whether they will affect a participant's ability to participate in the study procedures or will affect one or more outcome measures.
* Unable to distinguish colors used in Stroop task
* Use of oral corticosteroids
* Inability or unwillingness to withhold medication as detailed below, before each set of laboratory assessments:

  * Leukotriene Inhibitors - 2 days
  * Zyrtec - 5 days
  * Allegra/Claritin - 4 days
  * Antihistamines - 2 days
  * Nasal Steroids - 24h
  * Albuterol - 6 h
  * Inhaled corticosteroids - 12 h
* Use of >1000 mcg Fluticasone or equivalent ICS per day.
* Use of monoclonal antibody that targets eosinophils
* Concurrent medications other than for allergies/asthma (must be approved by Dr.)
* Current smoker or has a smoking history exceeding 5 pack-years within the last 10 years (i.e. someone who has been a non-smoker for 10 or more years can be enrolled)
* Significant previous training or significant current practice in meditation

  * Completed Mindfulness Based Stress Reduction (MBSR) in the past.
  * Current meditation practice. Judgment: Participants will be included or excluded at the PIs discretion due to wide variation in responses (e.g. 2 people answer yes, one practices mindfulness 2x/week for 2 years (exclude), the other attends regular religious services (include)).
* Significant daily practice with other mind-body techniques

  * Daily Yoga or Tai Chi Practice - exclude
  * Other daily practice - judgment.

Inclusion Criteria - MNP-NA:

* Able to provide valid informed consent to participate by signing/dating a consent form.
* Fluent English speaker
* MRI safe - Not excluded based on magnetic resonance Screening Form
* BMI under 35
* 25-65 years old
* Live within 50 miles of Madison, WI.
* Takes less than 30 minutes to fall asleep on average. Gets a good night of sleep regularly. Goes to bed before 12 a.m., able to sleep between 11 p.m. & 6 a.m. and sleeps >= 6 hours. (May be included at sleep doctor's discretion. In some cases, participants may not comply with these criteria but may be entirely safe to participate in the study. For example, a participant may indicate they do not get a good night of sleep due to a situational issue such as a waking baby or a pet as opposed to a chronic issue like insomnia. In these cases, there is no safety issue in having the participant included in the study)
* Participants assigned to HEP must have physician signature (on the Physician Authorization Form - PAF) indicating it is safe for them to participate in our interventions as some participant characteristics, such as a family history of coronary or atherosclerotic disease, represent risk factors that together may make the HEP intervention inadvisable; The process is consistent for ANY person who wishes to participate in any sort of physical activity class at the UW Health Research Park Clinic.
* Must be US citizen, green card holder or have an F-1 or J-1 visa. This is required in order to be able to pay participants.

Exclusion Criteria - MNP-NA:

* Pregnant, wanting to become pregnant, breast feeding or less than 6 months post-partum.
* Taking prescribed psychotropic or central nervous system altering medications (may be judged by PI in cases of periodic use (e.g. takes anti-anxiety med only when flying)
* History of a diagnosed Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder. Diagnosed episode of Major Depression unless it was more than 1 year ago. Diagnosed eating disorder or anxiety disorder unless it was more than 1 year ago.
* Excluded based upon the screening visit
* Some ongoing medical problems will be excluded based on team judgments about whether they will affect a participant's ability to participate in the study procedures or will affect one or more outcome measures.
* Unable to distinguish colors used in Stroop task
* Currently participating in another clinical trial
* Current diagnosis of asthma unless. History of asthma is not cause for exclusion.
* Taking prescribed sleeping medications (may be judged by sleep doctor in cases of periodic use (e.g. takes sleep med only when traveling internationally))
* Currently diagnosed sleep disorders. Past disorders are a judgment by a doctor from the sleep clinic.
* Regular night shift worker. (Participants may work periodic night shifts (e.g. one rotation per month) as long as they are able to sleep at normal times for the study)
* Epworth Sleepiness Scale - sleep lab will judge focusing on whether this a situational or chronic issue (e.g. dogs waking up vs. awake due to anxiety).
* Insomnia Severity Index - sleep lab will judge focusing on whether this a situational or chronic issue (e.g. dogs waking up vs. awake due to anxiety).
* STOP-BANG questionnaire - sleep lab will judge focusing on whether this is a situational or chronic issue (unless question 3 = yes in which case a score >3 will be excluded).
* Cigarette smoker unless willing to go without a cigarette for 4 hours or more.
* Traveled across more than 3 time zones in the three weeks prior to each study visit.
* Expert in physical activity (e.g. physical therapist, personal trainer), music (music therapist) or nutrition (nutritionist).
* Significant daily practice with physical activity as scored by the web screen.
* Significant previous training or significant current practice in meditation

  * Completed Mindfulness Based Stress Reduction (MBSR) in the past.
  * Current meditation practice. Judgment: Participants will be included or excluded at the PIs discretion due to wide variation in responses (e.g. 2 people answer yes, one practices mindfulness 2x/week for 2 years (exclude), the other attends regular religious services (include)).
* Significant daily practice with other mind-body techniques

  * Daily Yoga or Tai Chi Practice - exclude
  * Other daily practice - judgment.

Inclusion Criteria - LTM:

* Able to provide valid informed consent to participate by signing/dating a consent form.
* Fluent English speaker
* MRI safe - Not excluded based on magnetic resonance Screening Form
* BMI under 35
* 25-65 years old .
* Takes less than 30 minutes to fall asleep on average. Gets a good night of sleep regularly. Goes to bed before 12 a.m., able to sleep between 11 p.m. & 6 a.m. and sleeps >= 6 hours. Long-term practitioners may be judged on these last criteria because their sleep habits are sometimes very different than meditation naïve participants. (May be included at sleep doctor's discretion. In some cases, participants may not comply with these criteria but may be entirely safe to participate in the study. For example, a participant may indicate they do not get a good night of sleep due to a situational issue such as a waking baby or a pet as opposed to a chronic issue like insomnia. In these cases, there is no safety issue in having the participant included in the study)
* Meditation practice for a minimum of 5 years with an average practice of 200 minutes/week, that includes both mindfulness meditation and loving kindness and/or compassion meditation
* Significant retreat experience - a minimum of five weeks on retreat (with PI's discretion as financial means can make retreats impossible).
* Must be US citizen, green card holder or have an F-1 or J-1 visa. This is required in order to be able to pay participants.

Exclusion Criteria - LTM:

* Pregnant, wanting to become pregnant, breast feeding or less than 6 months post-partum.
* Taking prescribed psychotropic or central nervous system altering medications (may be judged by PI in cases of periodic use (e.g. takes anti-anxiety med only when flying)
* History of a diagnosed Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder. Diagnosed episode of Major Depression unless more than 1 year ago. Diagnosed eating disorder or anxiety disorder unless it was more than 1 year ago. Participants may be included with a history of these disorders with the PIs discretion.
* Excluded based upon the screening visit (Non-local LTMs will be excluded if they are not comfortable with the MRI however they may participate in the study if they are not comfortable with the electrical stimulation.)
* Some ongoing medical problems will be excluded based on team judgments about whether they will affect a participant's ability to participate in the study procedures or will affect one or more outcome measures.
* Unable to distinguish colors used in Stroop task
* Currently participating in another clinical trial
* Taking prescribed sleeping medications (may be judged by sleep doctor in cases of periodic use (e.g. takes sleep med only when traveling internationally))
* Currently diagnosed sleep disorders. Past disorders are a judgment by a doctor from the sleep clinic.
* Regular night shift worker. (Participants may work periodic night shifts (e.g. one rotation per month) as long as they are able to sleep at normal times for the study)
* Epworth Sleepiness Scale - sleep lab will judge focusing on whether this a situational or chronic issue (e.g. dogs waking up vs. awake due to anxiety).
* Insomnia Severity Index - sleep lab will judge focusing on whether this a situational or chronic issue (e.g. dogs waking up vs. awake due to anxiety).
* STOP-BANG questionnaire - sleep lab will judge focusing on whether this is a situational or chronic issue (unless question 3 = yes in which case a score >3 will be excluded).
* Cigarette smoker unless willing to go without a cigarette for 4 hours or more.
* Traveled across more than 3 time zones in the three weeks prior to each study visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2014-09; Primary Completion 2018-11 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Change in temporal dynamics of response to emotional anticipation task (fMRI) as a result of short term meditation practice OR 8 week training in meditation or health wellness interventions. | baseline, 3 months, 10 months
Change in slope measure of diurnal cortisol following a well-being intervention relative to baseline. | baseline (pre-intervention), 3 months (post-intervention), 10 months (follow-up)
Difference between groups (MBSR, WL) on change in lung function from pre-training to post-training | baseline (pre), 3 months (post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Davidson, PhD, Principal Investigator — UW-Madison, Center for Investigating Healthy Minds at the Waisman Center
Locations (4):
- United States (4):
  - UW Madison, Center for Investigating Healthy Minds at the Waisman Center, Madison, Wisconsin
  - UW-Madison, Asthma, Allergy and Pulmonary Research Center, Madison, Wisconsin
  - UW-Health Sports Medicine & Integrative Medicine Program, Madison, Wisconsin
  - Center for Sleep and Consciousness (and Wisconsin Sleep Clinic), Madison, Wisconsin

REFERENCES:
- [Derived] Higgins ET, Davidson RJ, Busse WW, Klaus DR, Bednarek GT, Goldman RI, Sachs J, Rosenkranz MA. Clinically relevant effects of Mindfulness-Based Stress Reduction in individuals with asthma. Brain Behav Immun Health. 2022 Sep 14;25:100509. doi: 10.1016/j.bbih.2022.100509. eCollection 2022 Nov. PMID 36177306